CLINICAL TRIAL: NCT02285660
Title: Evaluation of 4D-contrast Enhanced PET-CT in Tumour Volume Definition for Patients With Lung, Lower Oesophageal and Pancreatic Carcinomas.
Brief Title: Evaluation of 4D-contrast Enhanced PET-CT in Tumour Volume Definition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: The Leeds Teaching Hospitals Charitable Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: RD11/9711; 11/YH/0213 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-10-21; First posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Lung Carcinoma; Lower Oesophageal Carcinoma; Pancreatic Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Pancreatic Neoplasms

ARMS (2):
- Routine CT scan plus 4D PET-CT scan (Other)
  Interventions: Procedure: 4D PET-CT Scan
- Routine CT scan (Other)
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: 4D PET-CT Scan
  Arms: Routine CT scan plus 4D PET-CT scan
Other: No intervention
  Arms: Routine CT scan

SUMMARY:
The aim of high dose radiotherapy treatment is to deliver enough radiation to the tumour to kill all the cancer cells while at the same time giving a low dose of radiation to the normal parts of the body to reduce the side effects of treatment. This requires the cancer specialist to accurately identify the areas of cancer on a computed tomography (CT) scan. Positron emission tomography computed tomography (PETCT) scans use radioactive sugar that is injected into the patient. This sugar goes into cancer cells and shows up as a bright spot on the PET scan, allowing the doctors to see tumours more accurately. Some cancers move with breathing, for example lung, pancreas and oesophageal (or gullet) cancers. Fourdimensional CT scanning (4DCT) is a special type of CT scan that allows the motion of the tumour to be seen and measured accurately. This information can then be used to help ensure that the radiotherapy correctly treats the moving tumour.

The aim of this study is to see if there are possible benefits to combining PET with 4DCT to get a 4D PETCT scan for tumours that move with breathing. This study is divided into three cancer types; lung, lower oesophagus and pancreatic cancer.

First the investigators are going to test the use of 4D PETCT in the radiotherapy planning of these tumours to see if it helps the doctor to identify the cancer.

Secondly, the investigators are going to see if the 4D PETCT helps to show areas within the cancer that are potentially more active. This might then allow us to target a higher dose to these areas, which could potentially improve the chance of controlling and curing the cancer. Patients' standard treatment will not be altered by participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* WHO Performance status 02 (Appendix A)
* Histologically proven non small cell lung carcinoma, distal oesophageal carcinoma or pancreatic adenocarcinoma
* Clinical decision made to proceed with a course of radiotherapy of curative intent with or without concurrent chemotherapy
* Measurable primary tumour and/or locoregional metastatic lymph nodes on preradiotherapy imaging
* Able to provide fully informed written consent
* Able to lie flat for 1 hour
* Not be pregnant or breast feeding. Female patients of childbearing potential must agree to use effective contraception, be surgically sterile, or be postmenopausal.

Exclusion Criteria:

1. Hypersensitivity to Fluorine18 fludeoxyglucose (FDG)
2. Hypersensitivity to iodinated contrast media
3. Poorly controlled diabetes
4. Acute renal failure or moderate renal impairment (estimated glomerular filtration rate < 30 mL/min)
5. Claustrophobia precluding imaging
6. Uncontrolled pain
7. Urinary incontinence
8. Female patients must not be pregnant and if of child bearing age using adequate contraception
9. Breast feeding
10. Serious psychiatric comorbidity

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2011-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Whole body 4D PET-CT for improved Target Definition/Delineation (feasibility and benefit) (ability to identify the cancer and ability to show areas within the cancer that are potentially more active allowing target of higher dose to these areas) | Up to two hours
  To evaluate the feasibility and potential benefit of utilising 4D PET-CT for improved Target Definition/Delineation and to assess optimal segmentation of PET data

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Scarsbrook A, Ward G, Murray P, Goody R, Marshall K, McDermott G, Prestwich R, Radhakrishna G. Respiratory-gated (4D) contrast-enhanced FDG PET-CT for radiotherapy planning of lower oesophageal carcinoma: feasibility and impact on planning target volume. BMC Cancer. 2017 Oct 4;17(1):671. doi: 10.1186/s12885-017-3659-9. PMID 28978306